CLINICAL TRIAL: NCT03593369
Title: A Prospective Controlled Randomized Clinical Study Exploring The Evolution Of Wound Biomarkers With TWO Dispensing Schedules Of The KLOX LumiHeal Gel And The KT-L Lamp Versus Standard Of Care In Venous Leg Ulcers
Brief Title: Assessment of the Evolution of Wound Biomarkers in Venous Leg Ulcers Treated With KLOX Biophotonic System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CL-K1002-P013
Record Dates: First submitted 2018-07-10; First posted 2018-07-20 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- KLOX BioPhotonic System (single treatment)+SOC (Experimental): KLOX BioPhotonic System (LumiHeal Gel plus KLOX Multi-LED KT-L Lamp) will be administered twice weekly in association with SOC (10 patients)
  Interventions: Device: KLOX BioPhotonic System (single treatment)+SOC
- KLOX BioPhotonic System (consecutive treatments)+SOC (Experimental): KLOX BioPhotonic System (LumiHeal Gel plus KLOX Multi-LED KT-L Lamp) will be administered in two consecutive treatments (twice weekly on the first two weeks then once weekly) in association with SOC (10 patients)
  Interventions: Device: KLOX BioPhotonic System (consecutive treatments)+SOC
- Standard of Care (Active Comparator): SOC only (5 patients)
  Interventions: Other: Standard of Care (SOC)

INTERVENTIONS:
Device: KLOX BioPhotonic System (single treatment)+SOC — KLOX BioPhotonic system (composed of LumiHeal Gel and KT-L Lamp). In this study arm one treatment will be assessed - two visits per week.
  Standard of Care (SOC) for wound healing will be administered during the treatment and follow-up periods (20 weeks).
  Arms: KLOX BioPhotonic System (single treatment)+SOC
Device: KLOX BioPhotonic System (consecutive treatments)+SOC — In this study arm, two consecutive treatments during the same visit will be evaluated- two visits for the first two weeks, then one visit per week.
  Standard of Care (SOC) for wound healing will be administered during the treatment and follow-up periods (20 weeks).
  Arms: KLOX BioPhotonic System (consecutive treatments)+SOC
Other: Standard of Care (SOC) — Standard of Care (SOC) for wound healing will be administered during the treatment and follow-up periods (20 weeks).
  Arms: Standard of Care

SUMMARY:
The main purpose of the study is to evaluate the effect of KLOX BioPhotonic System (composed of KLOX LumiHeal Gel and KT-L Lamp) on the expression of wound biomarkers in the treatment of venous leg ulcers (VLU). Patients will be randomized in three groups, two different dispensing schedules of KLOX BioPhotonic System in addition to Standard of Care (SOC) will be used, and SOC alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 to 85 years of age, ambulatory or hospitalized patients;
2. Patient agrees to participate in protocol schedule of visits, including follow-up evaluations;
3. Patient to be enrolled must be able to adhere to the Standard of Care and to the treatments with the KLOX LumiHeal™ Gel and the KT-L Lamp described in the protocol;
4. Patient or an authorised person must be able to read and understand informed consent, and sign or delegate signature of the informed consent form;
5. Fitzpatrick skin type I to IV;
6. Proven venous leg ulcer, clinically defined and confirmed by duplex, refilling time or venous hypertension;
7. Ulcer to be treated must be measurable and with an area between 5 and 100 cm2 inclusively, with a maximum depth of 1 cm and maximum diameter less or equal to 10 cm;
8. If applicable, patients (male a female) must be willing to adhere to a medically-accepted birth control method (verified by the Investigator);
9. Stable wound surface area with an absolute change in wound area less than 30% as measured at Baseline Visit compared to the Screening Visit.

Exclusion Criteria:

1. Venous leg ulcer presents for less than 4 weeks or more than 18 months at Screening;
2. The patient has more than one ulcer in the treated leg and the ulcer(s) not being assessed are within 5 cm of the targeted ulcer;
3. The ulcer to be treated requires operative debridement or revascularization;
4. The ulcer has significant necrotic tissue, as defined by more than 20% of the ulcer area after debridement;
5. Major uncontrolled medical disorders such as serious cardiovascular, renal, liver or pulmonary disease, palliative care, or other chronic diseases such as lupus or sickle cell anemia;
6. Patient with known moderate to severe anemia;
7. Patient with history of malignancy within the wound or patient with prior diagnosis of malignant disease who is less than one year disease-free;
8. Patient who has experienced a hip fracture in the past 3 months;
9. Patient with known osteomyelitis or active cellulitis;
10. Patients who are immunosuppressed or on high dose of chronic steroid use (defined as oral dose of 7.5 mg or more of prednisone daily, or equivalent, for more than 28 days);
11. Patient with active wound infection or with systemic infection (the patient is however eligible for re-screening after the active wound infection or the systemic infection has subsided);
12. Successful revascularization surgery of the leg with the ulcer to be treated less than 8 weeks prior to Screening;
13. Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study, or participation within the past 60 days in another interventional wound healing clinical trial;
14. History of radiation therapy to the wound region;
15. Pregnancy, or breast feeding;
16. Patients with bleeding diathesis;
17. Patients on an uncontrolled anti-coagulation therapy;
18. The subject has any physical or psychiatric condition that, in the Investigator's opinion, would warrant exclusion from the study or prevent the subject from completing the study;
19. Concurrent disease or drugs known to induce severe photosensitivity of the skin, such as porphyria;
20. Patient has received biological-based therapy, skin grafts or Negative Pressure Wound Therapy in the ulcer to be treated within last 3 months prior to Baseline.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2018-07-09 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of biomarkers expression in biopsies and exudates of the venous leg ulcers. | Up to 20 weeks
  Comparison of the expression of biomarkers in biopsies and exudates of the venous leg ulcers in the three treatment groups.

SECONDARY OUTCOMES:
Adverse events, Serious adverse events, device incidents and compliance. | Up to 20 weeks
  Number of adverse events, serious adverse events, device incidents and missed treatment visits.

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Dini, MD, Principal Investigator — Azienda Ospedaliero, Universitaria Pisana
Locations (1):
- Clinica Dermatologica Azienda Ospedaliero-Universitaria Pisana, Pisa, Italy